CLINICAL TRIAL: NCT02313649
Title: Evaluation of ShearWave™ Elastography Performances for the Non-Invasive Assessment of Liver Fibrosis in Chinese Patients With Chronic Hepatitis B Infection
Brief Title: ShearWave™ Elastography to Assess Liver Fibrosis in Chinese Patients With Hepatitis B
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Responsible Party: Sponsor
Other Study IDs: LE2
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Liver Fibrosis
Keywords: liver; fibrosis; elastography; ShearWave Elastography; ultrasound
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate how liver stiffness measurements made with ShearWave™ Elastography (SWE) correspond with a biopsy result (currently the gold standard). The population that will be evaluated are Chinese patients infected with the Hepatitis B virus.

DETAILED DESCRIPTION:
Hepatitis B is becoming increasingly common. The liver becomes stiffer and this is called fibrosis. A non-invasive method to accurately stage fibrosis is necessary in order to begin the correct treatment. Currently, liver biopsy is used to do this, but there are many disadvantages with this technique.

ShearWave Elastography (SWE), available on the ultrasound machine Aixplorer®, is a non-invasive method to evaluate liver fibrosis.

This study will evaluate how liver stiffness measurements made with SWE correspond with a biopsy result (currently the gold standard).

The sensitivity, specificity, positive predictive value and negative predictive value of liver stiffness measurements with Aixplorer to evaluate the different stages of fibrosis will be analyzed.

Liver stiffness measurement made by the Aixplorer will also be compared to blood markers

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a liver ultrasound exam due to confirmed Hepatitis B infection ,
* Patients having reached the age of majority in China,
* Patients with a liver biopsy for histological evaluation of liver fibrosis, performed within 3 months after the SWE measurement date, and having the recommended quality criterion:

  * minimal length of biopsy samples of 15 mm, stored in paraffin
  * Minimal number of portal tracts of 6 per biopsy samples
* Patients of Chinese ethnic origin

Exclusion Criteria:

* Any patient presenting with combined etiologies of chronic liver diseases, including non-Hepatitis B viral infection（Hepatitis A, C, D, E, chronic alcoholic liver disease, hemochromatosis, autoimmune hepatitis, etc)
* History of antiviral therapy at any time
* Any patient presenting with a co-infection of HIV
* Any patient presenting with combined liver malignant tumor
* Previous liver transplantation
* Pregnant women
* Any patient with combined hepatic congestive condition such as Budd Chiari Syndrome, congestive heart failure, chronic constrictive pericarditis…
* Any patient combined with intrahepatic cholestasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with chronic viral hepatitis B admitted for the realization of an intercostal liver biopsy in defined investigator centers.
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Areas under the ROC curves for the ability of SWE measurements to predict at least significant fibrosis (Metavir F≥2), at least severe fibrosis (Metavir F≥3), and liver cirrhosis (Metavir F=4). | Within 12 months of the study start date
  This will be determined by histological examination of liver biopsy

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive values of SWE to predict at least significant fibrosis (Metavir F≥2), at least severe fibrosis (Metavir F≥3), and liver cirrhosis (Metavir F=4). | Within 12 months of the study start date
  This will be determined by histological examination of liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Principal Investigator — People's Liberation Army General（301）Hospital
Locations (15):
- China (15):
  - People's Liberation Army General（301）Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - 1st Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - 3rd Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - GuangZhou 8th People's Hospital, Guangzhou
  - 1st Affiliated Hospital, Haerbin Medical University, Haerbin
  - 1st Affiliated Hospital, ZheJiang University, Hangzhou
  - YunNan Province Second People's Hospital, Kunming
  - 2nd Affiliated Hospital, Lanzhou University, Lanzhou
  - Jiangsu Provincial Hospital, Nanjing
  - Shanghai 1st People's Hospital, Shanghai
  - Shengjing Hospital of Chinese Medical University, Shenyang
  - 1st Affiliated Hospital, XiAn Transportation University, Xi'an
  - Xijing Hospital, Xi'an
  - Isolation Hospital, HeNan Province, Zhengzhou

REFERENCES:
- [Derived] Wang K, Lu X, Zhou H, Gao Y, Zheng J, Tong M, Wu C, Liu C, Huang L, Jiang T, Meng F, Lu Y, Ai H, Xie XY, Yin LP, Liang P, Tian J, Zheng R. Deep learning Radiomics of shear wave elastography significantly improved diagnostic performance for assessing liver fibrosis in chronic hepatitis B: a prospective multicentre study. Gut. 2019 Apr;68(4):729-741. doi: 10.1136/gutjnl-2018-316204. Epub 2018 May 5. PMID 29730602